CLINICAL TRIAL: NCT00173394
Title: The Assessment of Mesothelin Antigen Specific Immunologic Assays in Ovarian Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700630
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2005-07

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; immunotherapy; mesothelin; normal volunteer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Ovarian cancer is the first in mortality rate of the gynecologic malignancies and the overall 5-year survival rate of ovarian cancer is only 20-30%. Besides, the incidence of ovarian cancer increased in recent years in Taiwan. Ovarian cancer is indeed a disease that should be respected, however, there has only been a little research done focusing on it in Taiwan. Patients with ovarian cancer who have stage I disease (localized to ovaries) after optimal surgical staging do not need any adjuvant therapy. In contrast, patients with disease spreading beyond the ovaries have median survival rates that decrease to < 10% for patients with bulky residual disease after surgery and treated with platinum-based combination chemotherapy. In developing effective therapy for ovarian cancer, there should be a distinction between preventative and therapeutic approaches. Immunoprevention will be developed for women who are at an increased risk for the development of ovarian cancer. In contrast, immunotherapy would be used as an adjuvant to surgery or in combination with chemotherapy or other biologics as chemoimmunotherapy or biochemoimmunotherapy. Mesothelin is expressed in some normal epithelial cells and is elevated in certain carcinomas. Mesothelin has been reported to be selectively overexpressed in most of the non-mucinous ovarian carcinomas. In addition, the specific epitopes of mesothelin in the HLA-A2 and A24 haplotype have been identified. It seems that mesothelin has the potential to be a target antigen for the immunotherapy of ovarian cancer.

So the investigators would like to provide this proposal to address the development of mesothelin -specific immunologic assays. There are two aims in this project:

1. to develop and utilize assays to measure cytotoxic T lymphocytes (CTLs) to mesothelin, and
2. to evaluate the mesothelin-specific immunologic responses between normal control and ovarian cancer patients.

DETAILED DESCRIPTION:
Incidence of Ovarian Cancer:

Ovarian cancer is the first in mortality rate of the gynecologic malignancies with an overall 5-year survival rate of only 20-30%. It became a more and more important disease in recent years and the incidence of ovarian cancer also increased in recent years in Taiwan. The lack of symptoms, difficulties in early diagnosis, insufficient accurate tumor markers, and lack of information about ovarian tumor biology contribute to the poor prognosis in ovarian cancer patients. The prognostic parameters for ovarian carcinomas are tumor stage, histologic subtype, degree of malignancy, and residual tumor after surgical treatment. However, these factors present an incomplete picture of the tumor biology of ovarian cancer and are frequently interrelated. Thus, the identification of new biologic factors predictive of individual disease course and prognosis would be extremely useful. From the above-mentioned data, ovarian cancer is indeed a disease that should be respected, however, there has only been a little research done focusing on it in Taiwan.

Treatment of Ovarian Cancer:

Epithelial Ovarian Cancer (EOC) and extraovarian Müllerian carcinoma are similar pathologic entities that share a preference for peritoneal cavity involvement. The spread pattern of these tumors presents a challenge and unique opportunities for immunotherapy. Patients with EOC who have stage I disease (localized to ovaries) after optimal surgical staging, have a 5-year survival rate of 90%, with no significant change at 10 years. In contrast, patients with spreading beyond the ovaries have median survival rates that decrease to < 10% for patients with bulky residual disease after surgery and treatment with platinum-based combination chemotherapy. A randomized trial of first-line chemotherapy in patients with EOC with residual masses larger than 1 cm after initial surgery, showed a median survival period of 38 months for cisplatin/paclitaxel, significantly greater than 24 months for the cisplatin/cytoxan treatment arm. In an interim analysis of an equivalency trial, survival after carboplatin/paclitaxel was not worse than cisplatin/paclitaxel. Even though early diagnosis is an important goal of ongoing clinical research efforts, it is unclear whether advanced EOC starts as a multicentric process involving the ovaries and the peritoneal surface. It is now established that hereditary factors contribute to the development of EOC. Germline BRCA1 and BRCA2 mutations account for approximately 10% of all EOC. In a woman with a BRCA 1 or 2 mutation, lifetime risk for ovarian cancer ranges from 16%-44%. With the commercial availability of genetic testing for BRCA1 and BRCA2, more women are being identified as being at high risk for ovarian cancer. There are no clear guidelines on cancer prevention for these individuals. Although prophylactic oophorectomy is a reasonable option for women who have completed childbearing, these women are still at risk for developing peritoneal cancer. Clearly, other options for prevention are needed.

Immunotherapy for Ovarian Cancer:

In developing effective immune-based strategies for EOC, there should be a distinction between preventative and therapeutic approaches. It is anticipated that immunoprevention (immunoprophylaxis) will be developed for women who are at an increased risk for the development of EOC. In contrast, immunotherapy would be used as an adjuvant to surgery or in combination with chemotherapy or other biologics as chemoimmunotherapy or biochemoimmunotherapy. Patients with undetectable disease after being restaged after chemotherapy could be considered for immunotherapy with the presumption that a majority does in fact have micrometastases. Development of effective immune-based concepts for prevention or treatment of EOC will require an understanding of tumor-immunology principles, mechanisms of action of the expanding array of immune modulating molecules, identification and characterization of tumor antigens, and determination of the microenvironment factors that could impact on the different immune-effector mechanisms. The clinical researcher has been provided with many immune directed agents, but progress on their integration into standard therapies has been somewhat slow.

Mesothelin:

Mesothelin is a 40-kDa glycosylphosphatidylinositol-linked glycoprotein. It is synthesized as a precursor of molecular mass 69 kDa, which then is proteolytically processed into an N terminal secreted form of molecular mass 30 kDa and a membrane-bound form of 40 kDa. In normal tissues, the expression of mesothelin has subsequently been shown to be largely restricted to mesothelial cells, although immunoreactivity has also been reported in epithelial cells of the trachea, tonsil, fallopian tube, and kidney. Hough et al. observed that mesothelin was over-expressed in ovarian carcinoma. It seems that mesothelin may be utilized as a tumor marker or target antigen for ovarian carcinoma.

Epitopes of Mesothelin for Human Haplotype:

The incidence of HLA-A2 haplotype is over 50% in the Western countries. The incidence of HLA-A2 and A24 haplotype is around 30% and 15% in Taiwan, respectively. The specific epitopes of the mesothelin in the HLA-A2 and A24 haplotype have been identified. There are Mesothelin aa20-28 (peptide SLLFLLFSL) and aa530-538 (peptide VLPLTVAEV) for the HLA-A2 haplotype. And Mesothelin aa435-443 (peptide FYPGYLCSL) and aa475-483 (peptide LYPKARLAF) are the epitopes of HLA-A24 haplotype.

Our research team has focused on the development of cancer vaccine and immunotherapy for several years. Our laboratory facilities have also been set up to evaluate the human immunologic assays for human papilloma virus type 16 E7 antigen by the grant supported from National Taiwan University Hospital. It is very important to set up various mesothelin-specific immunologic assays of human beings to evaluate the effect of cancer vaccine or immunotherapy for ovarian cancer in future clinical trials. So we would like to provide this proposal to address the development of mesothelin-specific immunologic assays in human beings. There are several aims in this project:

1. to develop and utilize assays to measure CTLs to mesothelin, and
2. to evaluate the mesothelin-specific immunologic responses between normal controls and ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and ovarian cancer patients will be enrolled from the investigators' department under the approval of the Institutional Review Board.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-08; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan